CLINICAL TRIAL: NCT04791410
Title: Clinical Study on the Efficacy of Microvascular Decompression in the Treatment of Neurogenic Hypertension
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Ruen, PekingUPH, Peking University People's Hospital
Other Study IDs: Neurogenic Hypertension
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Neurogenic Hypertension; Hypertension; Surgery
Keywords: neurogenic hypertension; microvascular decompression; hemifacial spasm
MeSH Terms: conditions — Hypertension; Hemifacial Spasm | interventions — Microvascular Decompression Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: patients who met the inclusion criteria were treated with RVLM decompression at the same time of facial nerve decompression.
  Interventions: Procedure: microvascular decompression
- control group: Patients who met the inclusion criteria were followed up for 3 months before surgery

INTERVENTIONS:
Procedure: microvascular decompression — Microvascular decompression of rostral ventrolateral medulla
  Groups: Experimental group

SUMMARY:
Hypertension has always been a threat to human health, so the prevention and treatment is of great significance. At present, the treatment of primary hypertension is mainly drug treatment, but many patients can not control their blood pressure in the normal range. Therefore, it is urgent to explore new and effective treatment methods.

Microvascular compression type of neurogenic hypertension is mainly due to abnormal tortuous vascular pulsatile compression of blood pressure center - rostral ventrolateral medulla (RVLM), resulting in the release of sympathetic active substances, leading to hypertension. The purpose of this study is to explore the efficacy and safety of microvascular decompression for hypertension in patients of hemifacial spasm complicated with hypertension, and to explore the common characteristics of patients with effective decompression.

The type of study design was prospective cohort study. According to certain inclusion and exclusion criteria, patients with RVLM compression were treated with RVLM decompression at the same time of facial nerve decompression. Patients who were followed up for 3 months were taken as control group, and the blood pressure of the two groups were measured after 3 months. The main outcome measure was 24-hour ambulatory systolic blood pressure change from baseline to 3 months.

DETAILED DESCRIPTION:
Research steps: If the patients with hemifacial spasm are complicated with hypertension and have the intention of surgical treatment, researchers would introduce the process, possible benefits and possible complications of the clinical trial in detail. Patients who agree to be enrolled and meet the inclusion conditions will sign the informed consent form.

The history of hypertension, the relationship between hypertension and hemifacial spasm, the highest blood pressure, oral medication, blood pressure maintenance, whether complicated with dyslipidemia, diabetes, smoking history, etc. Before operation, 24-hour ambulatory blood pressure monitoring was performed to record preoperative systolic blood pressure, diastolic blood pressure and heart rate. The measurement interval is automatically measured every 20 minutes in the daytime (8:00am ~ 10:00pm) and every 30 minutes at night (10:00pm ~ 8:00am). CBP was recorded in the morning (8:00-10:00 AM) before taking medication, and completed in the morning of 8:00-9:00 am the next day. The cuff was placed on the left upper arm. During the monitoring period, the patient was required to reduce the movement of the left upper arm as much as possible to avoid the cuff loosening or falling off, which would affect the measurement results. The record of effective monitoring times must be more than 80% and the covering time must be more than 20h, otherwise the measurement should be repeated. Patients should rest for at least 5 minutes before blood pressure measurement. The upper arm was placed at the heart level. Using OMRON electronic sphygmomanometer, the size of the cuff is suitable for the patient's upper arm circumference, covering at least 2 / 3 of the upper arm circumference. The blood pressure of both upper arms was measured, and the blood pressure of the higher side was taken as the criterion. Repeat the measurement at an interval of 1-2 min, and record the average value of the two readings. If the difference between the two readings of systolic or diastolic blood pressure is more than 5 mmHg, it should be measured again, and the average of the three readings should be taken as the baseline blood pressure measurement result.

Both the experimental group and the control group need to continue to take antihypertensive drugs orally, and the type and dose of drugs remain unchanged.

The experimental group was hospitalized and completed the corresponding hematology and imaging examination. The control group was followed up for 3 months, after the end of the follow-up can be hospitalized and improve the corresponding hematology and imaging examination. If the control group matched with the experimental group is excluded, the control group needs to be rematched. The experimental group received RVLM and (or) IX / X rez decompression at the same time of facial nerve decompression, while the control group received no operation.

Follow up: Patients should be followed up at 3 months. The following items were evaluated and recorded in CRF during follow-up

1. Physical examination;
2. Laboratory examination;
3. Vital signs (heart rate, respiration);
4. Ambulatory blood pressure examination
5. Office blood pressure
6. Antihypertensive medication: the patient's blood pressure and the use of antihypertensive drugs were closely monitored after the operation, and the adjustment time, the type and dosage of antihypertensive drugs after the adjustment were recorded when making adjustments according to the blood pressure and the cardiologist's suggestions.
7. Postoperative adverse reactions and duration / remission time: adverse reactions such as dizziness, headache, nausea and vomiting, tinnitus, hearing loss, diplopia, facial paralysis, drinking water cough and hoarseness. The above adverse reactions can be recovered in a few days after the operation. The duration of adverse reactions should be recorded and relieved in a few days after the operation.
8. Postoperative adverse events: such as patient death, acute cardiovascular events (such as cardiac arrest, ventricular fibrillation, myocardial infarction and hypertensive crisis), severe anesthesia or surgical complications (such as long-term mechanical ventilation due to inability to remove endotracheal intubation, pulmonary embolism, postoperative cerebral hemorrhage, severe intracranial infection), etc.

Statistical analysis: SPSS software was used to analyze the follow-up results of the intervention group and the control group. The general statistical test uses the two-sided test, and the one-sided test needs to be explained. P value less than or equal to 0.05 was used to judge whether the difference was statistically significant. The description of quantitative indicators will calculate the mean, standard deviation, median, quartile, minimum and maximum. The classification index is described by the number and percentage of cases. The demographic characteristics, general situation and baseline (before treatment) of the three groups were compared. Among them, t test was used for measurement data and chi square test was used for grade data. Binary logistic regression was used to further verify the influence of age, gender, side, BMI, family history of hypertension and changes of serum catecholamine on the effect of microvascular decompression in the treatment of neurogenic hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Preoperative MRI showed RVLM compression;
3. Primary hemifacial spasm without other secondary factors;
4. The office systolic blood pressure is higher than 140mmHg and the systolic blood pressure of ambulatory blood pressure is higher than 130mmHg;
5. Sign informed consent.

Exclusion Criteria:

1. Secondary hypertension, such as renal hypertension, vascular hypertension, etc;
2. No antihypertensive drugs were taken after admission and ambulatory blood pressure monitoring showed that the blood pressure was within the normal range;
3. Pregnancy plan or lactation period during pregnancy or within 2 years;
4. Patients with congestive heart failure (NYHA grade II-IV), myocardial infarction and unstable angina pectoris within 6 months before enrollment; patients with severe heart diseases, such as cardiogenic shock, arrhythmia requiring treatment, heart valve disease, etc;
5. Severe cerebrovascular diseases (hypertensive encephalopathy, cerebrovascular injury, stroke, transient ischemic attack, etc.) within 6 months before admission;
6. Patients with severe liver disease or dysfunction (ALT or AST > 2 times the upper limit of normal reference value);
7. Patients with renal impairment (male serum creatinine > 2.0mg/dl (176 μ mol / L), female serum creatinine > 1.8mg/dl (159 μ mol / L));
8. Other surgical contraindications, such as coagulation disorders, severe anemia, severe pulmonary infection, persistent state of asthma, upper respiratory tract infection, uncorrected respiratory failure, diabetic ketoacidosis, hepatic encephalopathy, hepatic coma, acute cerebral infarction, etc;
9. Type I diabetic patients; diabetic patients with poor glycemic control (FBG > 11.1 mmol / L) or type 2 diabetic patients with microalbuminuria;
10. Had Cushing's syndrome, coarctation of aorta, hyperthyroidism and other diseases in the past;
11. Patients can not cooperate with the test and follow-up, such as mental disorders, dementia, advanced tumor, etc;
12. If the antihypertensive drugs were adjusted within 2 weeks before admission, the patients were excluded or re enrolled after the blood pressure was stable for 2 weeks;
13. Preoperative anesthesia score ≥ grade III;
14. To screen those who participated in other clinical studies and used research drugs within 3 months before the trial, or planned to participate in other clinical studies during the trial period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemifacial spasm patients with hypertension in our center.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Decreased systolic blood pressure | 3 months
  After 3 months of treatment, 24 h ambulatory blood pressure was measured, systolic blood pressure was compared with baseline level, and the difference was calculated.

SECONDARY OUTCOMES:
Decreased diastolic blood pressure | 3 months
  After 3 months of treatment, 24 h ambulatory blood pressure was measured, diastolic blood pressure was compared with baseline level, and the difference was calculated.
Decreased office systolic blood pressure | 3 months
  After 3 months of treatment, office blood pressure was measured, systolic blood pressure was compared with baseline level, and the difference was calculated.
Decreased office diastolic blood pressure | 3 months
  After 3 months of treatment, office blood pressure was measured, diastolic blood pressure was compared with baseline level, and the difference was calculated.
The cure rate of hypertension 3 months after treatment | 3 months
effective rate of hypertension 3 months after treatment | 3 months

IPD SHARING:
Plan to Share IPD: No
All patient information is confidential.